CLINICAL TRIAL: NCT05203471
Title: Crossing the Divide: Piloting an Integrated Care Model to Bridge Rural-urban Healthcare Systems and Reduce Major Amputations Among Rural Patients With Diabetic Foot Ulcers
Brief Title: Crossing the Divide: Piloting Integrated Care to Reduce Amputations Among Rural Patients With Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-1338; R01DK132569-01 (NIH); Protocol Version 2/6/2025 (Other: UW Madison); SMPH/MEDICINE/INFECT DIS (Other: UW Madison)
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Foot; Diabetic Ulcer of Left Foot; Diabetic Ulcer of Right Foot; Amputation
Keywords: Multidisciplinary care; Integrated care; Rural disparities; Recruitment; Retention
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: This is an adaptive study design where recruitment and retention protocols are modified to improve involvement of rural study participants over three waves. Actively enrolled participants receive/ provide care for diabetic foot ulcers using a care algorithm and referral checklist. Results are compared to historical controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Historical controls (No Intervention): Patients with diabetic foot ulcers cared for by a primary care provider participating in the study prior to launching the integrated care intervention.
- Integrated care (Active Comparator): Patients with diabetic foot ulcers cared for by a primary care provider participating in the study after launching the integrated care intervention. Only patients who provide informed consent and enroll in the study will be treated with our integrated care model. All other patients with a participating primary care provider will be treated using a standard care model and will not be considered study participants.
  Interventions: Other: integrated care model

INTERVENTIONS:
Other: integrated care model — The investigators are piloting an integrated care model for rural patients with diabetic foot ulcers. The model uses two tools to promote collaboration between providers: a care algorithm and a referral checklist. The care algorithm will be used by rural primary care providers to guide integrated care addressing glycemic control, vascular disease, wound care, and infection. The referral checklist will be used by rural schedulers who place referrals to urban specialists. It prompts schedulers to fax appropriate supporting documents (e.g. notes, labs, vascular testing results) with the referral request.
  Arms: Integrated care

SUMMARY:
This project directly addresses the escalating national rate of major (above-ankle) amputations due to diabetic foot ulcers; it focuses on rural patients, who face 37% higher odds of major amputation compared to their urban counterparts. The project pilots the first integrated care model adapted to rural settings, an approach that has reduced major amputations in urban settings by approximately 40%. Pilot data will be used to improve recruitment and retention strategies and provide preliminary evidence of efficacy needed to conduct a robust, statewide efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare worker inclusion criteria:

  * Willing to provide informed consent
  * Willing to comply with study procedures
  * Rural providers (primary care physicians at the UW Health Belleville Family Medicine Clinic, diabetes and wound care specialists at Sauk Prairie Healthcare Diabetes and Wound Care Clinic) and schedulers placing referrals.
  * Employed at a participating clinic
  * For rural providers, confirm understanding that they will retain clinical discretion to deviate from the integrated care model if they think it would best serve the patient.
  * Available for the duration of the study
* Patient inclusion criteria:

  * Able and willing to provide informed consent.
  * Willing to comply with study procedures and be available for the duration of the study.
  * 18 years of age and older.
  * Patient with either type 1 or type 2 diabetes at a participating rural clinic.
  * Develops diabetic foot ulcer during enrollment period.

Exclusion Criteria:

* Healthcare worker exclusion criteria:

  * Insufficient overlap in work schedules between rural providers and scheduler based on clinic manager determination.
* Patient exclusion criteria:

  * receiving palliative care such that referral to urban centers for aggressive limb salvage would be inappropriate, as assessed by patient rural provider
  * insurance does not cover referral to the University of Wisconsin's specialty clinics
  * Not suitable for study participation due to other reasons at the discretion of the investigators.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Proportion of patients receiving guideline-concordant vascular and infectious disease care processes | up to 2 years and 3 months
  (proportion of integrated care patients receiving guideline-concordant vascular and infectious disease care within 3 months of their enrollment) minus (the proportion of historical patients receiving guideline-concordant vascular and infectious disease care within 3 months of participant enrollment)

SECONDARY OUTCOMES:
Proportion of patients undergoing amputation | up to 2 years and 3 months
  (proportion of integrated care patients undergoing amputation within 3 months of their enrollment) minus (proportion of historical patients undergoing amputation within 3 months of their enrollment), where amputation is defined as major or minor amputation of the ipsilateral lower extremity to the index ulcer

OTHER OUTCOMES:
Patient recruitment rate | up to 2 years and 3 months
  Number of patients who enrolled in the study divided by the number of patients the study team attempted to contact for study recruitment
Patient retention rate | up to 2 years and 3 months
  Number of patients who completed the 3-month follow-up telephone call divided by the number of patients who enrolled in the study

CONTACTS AND LOCATIONS:
Overall Officials: Meghan B Brennan, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the study, after de-identification will be available to researchers for independent verification of study outcomes or to conduct subsequent clinical research, whose proposed use of the data has been approved by an independent review committee identified for this purpose.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months after publication of primary outcomes and ending 5 years after that date.
Access Criteria: Proposals should be directed to the PI, Dr. Meghan Brennan (mbbrennan@medicine.wisc.edu). If approved after review by regulatory counsel, requestors will enter into a formal data sharing agreement. Data will be shared via encrypted single-user file transmission protocol.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT05203471/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT05203471/ICF_000.pdf